CLINICAL TRIAL: NCT02989012
Title: Phase IIaTrials of GanMaoKangNing Granules
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dalian Zhen-Ao Bio-Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DalianZhen-Ao
Record Dates: First submitted 2016-11-30; First posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-11

CONDITIONS: Epidemic Influenza
MeSH Terms: interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drugs for experimental group (Experimental): GanMaoKangNing Granules， blunted by boiled water , 3 times a day, 2 bags each time, for a course of five days(During experiments, The condition of the subjects sicker or complications, Whether need to change or increase the treatment measures were determined by the researchers ,Stop using the medicine , completion of the relevant inspection and evaluation after medication,Quit the test,the case according to the invalid qualified cases statistics.); Analogous Oseltamivir Phosphate Capsules,take oral,2 times a day,1 capsule each time, for a course of five days(During experiments, The condition of the subjects sicker or complications, Whether need to change or increase the treatment measures were determined by the researchers ,Stop using the medicine , completion of the relevant inspection and evaluation after medication,Quit the test,the case according to the invalid qualified cases statistics.).
  Interventions: Drug: GanMaoKangNing Granules; Drug: Analogous Oseltamivir Phosphate Capsules
- Drugs for control group (Sham Comparator): Oseltamivir Phosphate Capsules ,take oral,2 times a day,1 capsule each time, for a course of five days(During experiments, The condition of the subjects sicker or complications, Whether need to change or increase the treatment measures were determined by the researchers ,Stop using the medicine , completion of the relevant inspection and evaluation after medication,Quit the test,the case according to the invalid qualified cases statistics.); Analogous GanMaoKangNing Granules, blunted by boiled water , 3 times a day, 2 bags each time, for a course of five days(During experiments, The condition of the subjects sicker or complications, Whether need to change or increase the treatment measures were determined by the researchers ,Stop using the medicine , completion of the relevant inspection and evaluation after medication,Quit the test,the case according to the invalid qualified cases statistics.).
  Interventions: Drug: Oseltamivir Phosphate Capsules; Drug: Analogous GanMaoKangNing Granules

INTERVENTIONS:
Drug: GanMaoKangNing Granules — 3 times a day, 2 bags each time.
  Arms: Drugs for experimental group
Drug: Analogous Oseltamivir Phosphate Capsules — 2 times a day,1 capsule each time.
  Arms: Drugs for experimental group
Drug: Oseltamivir Phosphate Capsules — 2 times a day,1 capsule each time.
  Arms: Drugs for control group
Drug: Analogous GanMaoKangNing Granules — 3 times a day, 2 bags each time.
  Arms: Drugs for control group

SUMMARY:
Randomized, double-blind, double- simulation, positive drug-and-Placebo-Controlled, multicenter, phase IIa clinical trials Study about GanMaoKangNing Granules in improving the symptoms of influenza.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent;
* Male and female patients aged between 18 and 65 years old , there is no limit on the gender;
* In line with the diagnostic criteria for pandemic influenza;
* Duration less than 48 (Duration is defined as the time from onset to test drugs for the first time before, the onset time pointed out that now the axillary temperature 38.0 ℃, headache, muscle or joint pain, chills, fatigue, cough, sore throat and a stuffy nose eight any flu symptoms and signs in time);
* The axillary temperature is 38.0 ℃ or higher;
* Nose and throat swabs rapid virus antigen test result is positive.

Exclusion Criteria:

* Severe influenza and of patients with complications of influenza.
* With the following any severe risk factors:

A. With chronic respiratory diseases such as bronchial asthma, chronic obstructive pulmonary disease (copd), etc.

B. with chronic diseases of the cardiovascular system, such as congestive heart failure, high blood pressure.

C. with chronic metabolic and endocrine system diseases, such as poorly controlled diabetes (HbA1c 7.0% or higher).

D. with chronic kidney disease, chronic liver disease, blood system diseases, neurological and neuromuscular diseases (such as epilepsy, cognitive impairment, etc.).

E. A weakened immune system, such as long-term use of immunosuppressive agents, HIV infection or tumor.

F. Under the age of 19, long-term aspirin use. G. The obese (BMI BMI > 30).

* With influenza complications, such as secondary bacterial pneumonia and other pathogenic bacteria and other viral pneumonia caused by pneumonia.
* A history of peptic ulcer disease or gastrointestinal bleeding.
* Into the group received within 48 h before flu antiviral treatment.
* Into the group of 12 months before been vaccinated against the flu.
* Into the group used within 2 weeks before the monoamine oxidase inhibitors.
* Blood leukocyte count > 10.0 x 109 / L, neutrophils ratio > 80%, or the need for systemic antibiotic therapy.
* For GanMaoKangNing Granules, Oseltamivir Phosphate Capsules, Acetaminophen Tablets, Dextromethorphan Hydrobromide Capsule, GanMaoKangNing Granules simulation agent or Oseltamivir Phosphate Capsules simulation agent composition of allergy, or allergic constitution.
* Aminotransferase (AST/SGOT) or alanine aminotransferase (ALT/SGPT) ≥ 1.5 x Upper Limit Normal (ULN)， Scr > Upper Limit Normal (ULN).
* Doubt or does have a history of alcohol or drug abuse.
* Pregnancy (defined as the pregnancy test positive), nursing mothers, or past in family planning.
* For nearly three months participated in other clinical trials of patients.
* Researchers think not appropriate to participate in this clinical subjects.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Primary Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Flu recovery time | six days
  All the time needed for symptoms eased that from medication to fever and headache, muscle joint pain, chills, fatigue, cough, sore throat and a stuffy nose.

SECONDARY OUTCOMES:
Single symptom remission rate | six days
  After the medication and three days later, The proportion of each individual symptoms of subjects which include of headache, muscle joint pain, chills, fatigue, cough, sore throat and a stuffy nose.
  Symptoms defined as symptom scores dropped to 0 or 1 minute, and maintain for 24 h or more.
The antifebrile effect | six days
  Antifebrile rate: After the medication and three days later, the percentage of Body temperature returned to normal subjects (the axillary temperature < 37.1 ℃, and maintain of 24 h or more time).
  Medicine antifebrile time (h) : Medication for the first time to the axillary temperature < 37.1 ℃, and maintain of 24 h or more time.

OTHER OUTCOMES:
The conditions of drug utilization of the antipyretic and some cough medicine | six days
  Including acetaminophen tablets and capsule of dextromethorphan hydrobromide usage rate and dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital of Traditional Chinese Medicine Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- See also: WHO. Influenza（Seasonal）[EB/OL].[2015-12-31] — http://www.who.int/mediacentre/factsheets/fs211/en/.